CLINICAL TRIAL: NCT05316207
Title: Investigation of the Effect of Tele-Nursing on Anxiety And Complications in Patients With Open Heart Surgery
Brief Title: Tele-Nursing Follow-Up After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Kadiriye Pehlivan, Principal Investigator, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TelenursingOHS
Record Dates: First submitted 2022-03-14; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Open Heart Surgery; Tele-nursing
Keywords: Anxiety; Complication; Readmission; Hospitalization
MeSH Terms: conditions — Anxiety Disorders | interventions — Telenursing

STUDY DESIGN:
Who Masked: Participant
Masking Description: Intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): IG was formed from 40 patients who received routine care, treatment and education services of the clinic after open heart surgery, and whose routine controls were determined by the randomization method. The patients in the IG would call by the researcher at least four times, at the end of the first, second, third and fourth weeks after discharge, to provide education and counseling via tele-nursing. In these phone calls, the current problems of the patient, if any, and the issues that should be paid attention to during the home care process after open heart surgery were explained.It was stated that, unlike the patients in CG, patients in IG would be called by the researcher at least four times at the end of the first, second, third and fourth weeks after discharge to provide education and counseling via tele-nursing.
  Interventions: Other: Telenursing
- Control Group (No Intervention): The patients in the CG were formed from 40 patients who received routine care, treatment and education services of the clinic after open heart surgery, and who were determined by the randomization method, whose routine controls were made after discharge. No application was made to the patients in the CG by the researcher within the scope of the study. However, the researcher gave the phone number to the patients in the CG in terms of their right to receive ethical and professional care, and it was stated that they could call between 10:00 and 22:00 if needed. The reasons for calling the investigator from the CG were recorded .

INTERVENTIONS:
Other: Telenursing — From the end of the first week after discharge to the end of the first month, patients were counseled over the phone during the home process. Complications were followed up.
  Arms: Intervention Group

SUMMARY:
Introduction: Failure to follow-up patients by healthcare professionals after discharge may increase the development of anxiety and complications in patients.

Aim: The aim of this study is to determine the effects of tele-nursing method to patients who have undergone Open Heart Surgery (OHS) after discharge on anxiety and some other complications.

Material and Methods:This quasi-experimental randomized controlled study, which was conducted in a private hospital between November 2020 and April 2021, included 75 patients, 38 from the Intervention (IG) and 37 from the Control Group (KG). IG and CG patients were provided routine treatment and care. In addition to the IG, training and counselling were provided at least four times by phone calls between the first week after discharge and the end of the first month. Descriptive Form and State-Trait Anxiety Inventory (STAI-S and T) were administered to all patients before discharge, and STAI-S was administered at the end of the first month after discharge. Post-discharge complications were evaluated by medical doctor in both groups. These data, number of hospitalization and readmission rates were obtained from hospital records.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years and older,
* Able to speak and understand Turkish,
* Without hearing, comprehension, vision and speech problems,
* Open heart surgery for the first time,
* Those who were not diagnosed with depression or anxiety disorder before surgery and didn't use medication for this purpose,
* Having a mobile phone that can take photos by herself/himself or her/his attendants,
* No serious complications to delay hospital discharge,
* Patients who volunteered to participate were included in the study.

Exclusion Criteria:

Patients who wished to withdraw from the study after volunteering were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Determination of change in anxiety levels between groups before discharge and one month after discharge | State and trait anxiety levels were measured 72 hours before discharge for all participants who met the inclusion criteria.State anxiety levels of all participants were measured one month after discharge.
  Anxiety levels of all participants who met the inclusion criteria were measured using the state and trait anxiety scale in the pre-test. At the end of the first week after discharge, the intervention was started for the patients in the study group and the intervention was completed at the end of the first month after discharge. One month after discharge, the state anxiety levels were measured again with the state anxiety scale.

SECONDARY OUTCOMES:
Rates of Complication Development | Complications developed in both groups were recorded at the end of the first week and the end of the fourth week after discharge.
  The rate of total hospitalization before and after the intervention, the rate of admission to the hospital for examination, leg incision infection, effusion, chest incision infection and other complications that may occur within one month after discharge, according to the groups

CONTACTS AND LOCATIONS:
Overall Officials: Kadiriye Pehlivan, MSc RN, Principal Investigator — Hasan Kalyoncu University; Ayla Yava, Prof, RN, Study Director — Hasan Kalyoncu Üni̇versi̇tesi̇ University
Locations (1):
- Medical Park Hospital, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No